CLINICAL TRIAL: NCT02206256
Title: Omega-3 Fatty Acids in Bariatric Gastric Bypass Surgery: Effect on Liver Volume, Immune Response and Erythrocyte Function
Acronym: OLIVIER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, Alexander P.J. Houdijk, Dr., Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL47021.029.13
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low calorie diet (Active Comparator): Low calorie diet 2 weeks pre-operatively
  Interventions: Behavioral: Low calorie diet
- Omega-3 fatty acid capsules (Active Comparator): 2 times a day 1 capsule for 4 weeks before gastric bypass surgery
  Interventions: Drug: Omega-3 fatty acid capsules

INTERVENTIONS:
Drug: Omega-3 fatty acid capsules — 2 times a day 1 capsule for 4 weeks before gastric bypass surgery
  Other Names: purified fish oil; omega-3 fatty acids; eicosapentoenoic acid (EPA); docosahexaenoic acid (DHA)
  Arms: Omega-3 fatty acid capsules
Behavioral: Low calorie diet — A low calorie diet of 600 kcal/day during 2 weeks, using Modifast or an adjusted normal diet.
  Arms: Low calorie diet

SUMMARY:
Gastric bypass surgery is the gold standard in bariatric surgery and is a successful method to reduce weight in morbidly obese subjects. Patients qualified for gastric bypass surgery are routinely pre-treated with a low calorie diet in order to reduce liver volume and to facilitate the approach of the gastro-oesophageal junction. Pre-treatment with omega-3 fatty acids has similar effects on liver volume, but a prospective comparison of both treatments has not been performed yet. Morbidly obese patients respond differently to surgical stress, due to a number of factors. First, obesity is associated with a low-grade inflammatory state induced by an increased amount of macrophages in adipose tissue. This state is associated with higher levels of pro-inflammatory cytokines in serum and with a less adequate immune response to infections. Second, obesity is associated with an altered cortisol metabolism possibly related to adrenal insufficiency. This could play an important role in the altered response to surgical stress and postoperative complications in obese subjects. Third, obesity is associated with altered erythrocyte function, including decreased erythrocyte deformability and increased aggregation, factors contributing to an impaired microcirculation.

This study has a number of different aims. First, we will compare pre-treatment with the standard low calorie diet with omega-3 fatty acids on liver volume in patients qualified for gastric bypass surgery because of morbid obesity. Second, we will investigate the effect of omega-3 fatty acids on immune function, the low-inflammatory state of adipose tissue, the stress response of obese subjects before and erythrocyte function. Third, we will investigate the effect of gastric bypass surgery by comparing values before surgery with values on the first postoperative day and 6 months after surgery regarding to immunological parameters, stress response and erythrocyte function.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing laparoscopic gastric bypass surgery because of morbid obesity
* Age between 18 and 65 years
* Able to fit in the MRI
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus type 1
* Current history of inflammatory, infectious or malignant disease
* Daily use of anti-inflammatory drugs
* Contra-indications for MRI imaging
* Contra-indications for the use of omega-3 fatty acids

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Liver volume | baseline, after treatment
  liver volume of the left hepatic lobe measured by MRI

SECONDARY OUTCOMES:
Peri-operative ex vivo LPS stimulated cytokine production capacity | baseline, operation day, postoperative day 1, follow up 6 months
  IL-6, IL-10, TNF-alpha
Macrophage infiltration in omentum fat biopsies | Biopsies during gastric bypass surgery
Erythrocyte function | baseline, day of surgery, postoperative day 1, follow up 6 months
  Measurement of erythrocyte deformability and aggregation with LORRCA (laser-assisted optical rotational red cell analyzer)
Cortisol response | baseline, operation day, postoperative day 1, follow up 6 months
  ACTH stimulation test
Serum parameters of inflammatory response | baseline, operation day, postoperative day 1, follow up 6 months
  IL-6, IL-10, TNF-alpha and C-reactive protein
Assessment of the approach of the gastro-oesophageal junction | During gastric bypass surgery
  Surgeons fill out a questionnaire after the gastric bypass surgery
Patient satisfaction with intervention | After the pre-operative treatment
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: A.P.J. Houdijk, Dr., Principal Investigator — Rode Kruis Ziekenhuis, Medisch Centrum Alkmaar
Locations (1):
- Rode Kruis Ziekenhuis, Beverwijk, North Holland, Netherlands

REFERENCES:
- [Derived] Bakker N, van den Helder RS, Geenen RWF, Hunfeld MA, Cense HA, Demirkiran A, Houdijk APJ. Four Weeks of Preoperative Omega-3 Fatty Acids Reduce Liver Volume: a Randomised Controlled Trial. Obes Surg. 2019 Jul;29(7):2037-2044. doi: 10.1007/s11695-019-03814-7. PMID 30888593